CLINICAL TRIAL: NCT02567461
Title: Effects of Edoxaban on the Cellular and Protein Phase of Coagulation in Patients With Coronary Artery Disease on Dual Antiplatelet Therapy With Aspirin and Clopidogrel (EDOX-APT): A Prospective Randomized Study
Brief Title: Edoxaban in Patients With Coronary Artery Disease on Dual Antiplatelet Therapy With Aspirin and Clopidogrel
Acronym: EDOX-APT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS DSI001
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: dual antiplatelet therapy; clopidogrel; aspirin; edoxaban
MeSH Terms: conditions — Coronary Artery Disease | interventions — edoxaban; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DAPT plus high-dose edoxaban (Experimental): High-dose edoxaban will be represented by edoxaban 60mg od, which will be reduced to 30mg od in patients with ClCr ≤50mL/min.
  Interventions: Drug: Edoxaban 60 mg; Drug: Clopidogrel 75 mg; Drug: Aspirin 81 mg
- DAPT plus low-dose edoxaban (Experimental): Low-dose edoxaban will be defined as edoxaban 30mg od, which will be reduced to 15mg od in patients with ClCr ≤50mL/min.
  Interventions: Drug: Edoxaban 30 mg; Drug: Clopidogrel 75 mg; Drug: Aspirin 81 mg
- DAPT (Active Comparator): Aspirin 81 mg od plus clopidogrel 75 mg od
  Interventions: Drug: Clopidogrel 75 mg; Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Edoxaban 60 mg — Patients will receive randomized treatment for 10±2 days, in order to achieve steady-state anticoagulant effects. Afterwards, patients randomized to any of the edoxaban groups (arms 1 and 2) will stop aspirin therapy. Study treatment will be administered for other 10±2 days.
  Other Names: Savaysa
  Arms: DAPT plus high-dose edoxaban
Drug: Edoxaban 30 mg — Patients will receive randomized treatment for 10±2 days, in order to achieve steady-state anticoagulant effects. Afterwards, patients randomized to any of the edoxaban groups (arms 1 and 2) will stop aspirin therapy. Study treatment will be administered for other 10±2 days.
  Other Names: Savaysa
  Arms: DAPT plus low-dose edoxaban
Drug: Clopidogrel 75 mg — Patients will receive randomized treatment for 10±2 days, in order to achieve steady-state anticoagulant effects. Afterwards, patients randomized to any of the edoxaban groups (arms 1 and 2) will stop aspirin therapy. Study treatment will be administered for other 10±2 days.
  Other Names: Plavix
Drug: Aspirin 81 mg — Patients will receive randomized treatment for 10±2 days, in order to achieve steady-state anticoagulant effects. Afterwards, patients randomized to any of the edoxaban groups (arms 1 and 2) will stop aspirin therapy. Study treatment will be administered for other 10±2 days.
  Other Names: ASA

SUMMARY:
It is not uncommon that patients requiring dual antiplatelet therapy (DAPT) also need to be treated with oral anticoagulant therapy, such as those with atrial fibrillation (AF). Warfarin and clopidogrel are still the most widely utilized oral anticoagulant and P2Y12 receptor inhibitor, respectively. However, over the past years, several non-vitamin K antagonist oral anticoagulants, including edoxaban, have been studied in the setting of AF showing encouraging safety and efficacy profiles as compared with warfarin. However, the effects of edoxaban in combination with DAPT in the setting of patients with coronary artery disease (CAD) are unexplored. Moreover, the role of edoxaban as part of a dual antithrombotic treatment strategy, including clopidogrel and stopping aspirin, represents another important area of clinical interest. This investigation is a prospective, randomized, parallel-design, open label, pharmacodynamic study conducted in patients with CAD on DAPT with aspirin and clopidogrel testing two different edoxaban dosing regimens in addition to DAPT with aspirin and clopidogrel, as well as in combination with clopidogrel only (after stopping aspirin).

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 receptor antagonist is pivotal for the treatment of patients with coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI) and in patents following an acute coronary syndrome (ACS). Importantly, it is not uncommon that patients requiring DAPT also need to be treated with oral anticoagulant therapy, such as those with atrial fibrillation (AF). Warfarin and clopidogrel are still the most widely utilized oral anticoagulant and P2Y12 receptor inhibitor, respectively. However, this treatment regimen has shown to be associated with an increased risk of bleeding, as well as ischemic complications. Over the past years, several non-vitamin K antagonist oral anticoagulants (NOACs), including edoxaban, have been studied in the setting of AF showing encouraging safety and efficacy profiles as compared with warfarin. In the phase III ENGAGE AF-TIMI 48 trial, edoxaban (60mg or 30mg once/daily) was non-inferior to warfarin with respect to the prevention of stroke or systemic embolism and was associated with significantly lower rates of bleeding and death from cardiovascular causes, in patients with AF. However, the effects of edoxaban in combination with DAPT in the setting of patients with CAD are unexplored. This may indeed represent a limitation for the uptake of edoxaban in modern day clinical practice where ~10% of patients with AF also have CAD requiring PCI and thus may require triple antithrombotic therapy. Moreover, the role of edoxaban as part of a dual antithrombotic treatment strategy, including clopidogrel and stopping aspirin, represents another important area of clinical interest as it has the potential reduce the risk of bleeding while preserving protection from ischemic events. This investigation is a prospective, randomized, parallel-design, open label, pharmacodynamic study conducted in patients with CAD on DAPT with aspirin and clopidogrel testing two different edoxaban dosing regimens (60mg or 30mg once/daily) in addition to DAPT with aspirin and clopidogrel, as well as in combination with clopidogrel only (after stopping aspirin).

ELIGIBILITY:
Inclusion criteria:

1. Patients with angiographically documented CAD (previous PCI or ACS).
2. On DAPT with low-dose aspirin (81mg od) and clopidogrel for at least 30 days as per standard-of-care.
3. Age above 18.

Exclusion criteria:

1. Active pathological bleeding, history of clinically significant bleeding events, or deemed at increased risk of bleeding.
2. CrCL <15mL/min
3. Any clinical indication to be on anticoagulant therapy
4. Acute coronary events in the past 90 days
5. Prior hemorrhagic stroke or intracranial hemorrhage
6. Ischemic stroke/transient ischemic attack in the past 6 months
7. Chronic use of nonsteroidal anti-inflammatory drugs
8. On treatment with rifampin (induce or P-gp transporter)
9. Known moderate or severe hepatic impairment (Child-Pugh B and C).
10. On treatment with any antiplatelet agent other than aspirin and clopidogrel in the past 30 days.
11. Platelet count <80x106/mL
12. Hemoglobin <10g/dL
13. Hemodynamic instability
14. Pregnant females [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Thrombin-activated clot strength with or without edoxaban | 10 days
  Comparison of thrombin-activated clot strength measured by TEG 6s system system between patients on DAPT plus high-dose edoxaban and patients on DAPT

SECONDARY OUTCOMES:
Thrombin-activated clot strength with or without aspirin | 10 days
  Comparison of thrombin-activated clot strength measured by TEG 6s system system between patients on DAPT plus high-dose edoxaban and patients on clopidogrel plus high-dose edoxaban

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No